CLINICAL TRIAL: NCT00516737
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Factorial Design Clinical Trial to Study the Efficacy and Safety of MK0462 / Rizatriptan 10 mg for the Early Treatment of Acute Migraine
Brief Title: Study to Test Rizatriptan in the Early Treatment of Acute Migraine (0462-081)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-081; 2007_547
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Results first posted 2009-04-14 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2022-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Active Drug
  Interventions: Drug: Comparator: rizatriptan benzoate
- 2 (Placebo Comparator): Matching Pbo Comparator
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: rizatriptan benzoate — Rizatriptan 10 mg Orally Disintegrating Tablet (ODT); one dose, treatment of a single migraine attack
  Other Names: MK0462
  Arms: 1
Drug: Comparator: Placebo — Matching placebo; one dose, treatment of a single migraine attack
  Arms: 2

SUMMARY:
The purpose of this study is to test the effectiveness of rizatriptan benzoate in the early treatment of an acute migraine attack.

ELIGIBILITY:
Inclusion Criteria:

* Greater than one year history of migraine
* Attacks typically mild when they begin and progress to moderate or severe
* Experience 1-4 migraine attacks per month

Exclusion Criteria:

* More than 15 headache days per month
* Heart disease
* Uncontrolled high blood pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2007-10-03 (Actual); Primary Completion 2008-04-08 (Actual); Study Completion 2008-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cady RK, Martin VT, Geraud G, Rodgers A, Zhang Y, Ho AP, Hustad CM, Ho TP, Connor KM, Ramsey KE. Rizatriptan 10-mg ODT for early treatment of migraine and impact of migraine education on treatment response. Headache. 2009 May;49(5):687-96. doi: 10.1111/j.1526-4610.2009.01412.x. PMID 19472447

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III First Patient In: 03-October-2007 Last Patient Last Visit: 08-April-2008 13 outpatient centers worldwide (10 United States, 3 Germany)
Pre-assignment Details: Participants were assessed, using the protocol inclusion and exclusion criteria, at Visit 1, and if eligible were randomized at that same visit.
Groups:
- Rizatriptan 10 mg ODT: Rizatriptan 10 mg Orally Disintegrating Tablet (ODT); one dose, treatment of a single migraine attack
- Placebo: Matching placebo; one dose, treatment of a single migraine attack
Period: Overall Study
Arm/Group | Rizatriptan 10 mg ODT | Placebo
Started | 103 | 104
Completed | 92 | 96
Not Completed | 11 | 8
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Qualifying Event | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rizatriptan 10 mg ODT | Placebo | Total
Number analyzed (Participants) | 103 | 104 | 207
Age, Continuous [Mean (Full Range); unit: years] | 41 [19 to 69] | 44 [18 to 66] | 42.5 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 96 | 186
  Male | 13 | 8 | 21
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 4 | 3 | 7
  White | 95 | 100 | 195
  Asian | 2 | 1 | 3
  Multi-Racial | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Pain Free at 2 Hours Post-Dose
Description: Pain severity was rated by the participants in a paper diary. Pain severity rating scale: 0 (no pain), 1 (mild), 2 (moderate), or 3 (severe). Pain free = rating of 0 (no pain) at 2 hours post-dose.
Time Frame: 2 hours post-dose
Population: Full Analysis Set (FAS): The FAS population includes all randomized participants who have at least one assessment within 2 hours post-dose (i.e., after baseline assessment).
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg ODT | Placebo
Number analyzed (Participants) | 92 | 96
Participants | 61 | 27

2. Secondary Outcome: Number of Participants With 24-Hour Sustained Pain Freedom
Description: 24-hour sustained pain freedom (defined as pain freedom from 2 to 24 hours post-dose and no use of rescue medication). Participants assessed pain severity and use of rescue medication on a paper diary.
Time Frame: 24 hours post-dose
Population: The FAS population was used for this secondary variable of 24-hour sustained pain freedom, unless participants were otherwise identified as non-responders for this endpoint (i.e., took rescue up to 24 hours post-dose or were not pain free at 2 hours post-dose). To be included, participants must have also had a non-missing 24-hour assessment.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg ODT | Placebo
Number analyzed (Participants) | 92 | 96
Participants | 48 | 17

3. Secondary Outcome: Number of Participants With no Rescue Use up to 24 Hours Post-Dose
Description: Participants recorded use of any rescue medication up to 24 hours after dosing with study medication on a paper diary.
Time Frame: 24 hours post-dose
Population: The FAS population included all randomized and treated participants.
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg ODT | Placebo
Number analyzed (Participants) | 92 | 96
Participants | 61 | 32

4. Secondary Outcome: Number of Participants With Absence of Photophobia at 2 Hours Post-dose
Description: Absence or presence of photophobia was recorded by the participants on a paper diary. Absence is defined as no photophobia at 2 hours post-dose.
Time Frame: 2 hours post-dose
Population: The FAS population included all randomized participants who had at least one assessment within 2 hours post-dose (i.e., after baseline assessment).
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg ODT | Placebo
Number analyzed (Participants) | 92 | 96
Participants | 69 | 43

5. Secondary Outcome: Number of Participants With Absence of Phonophobia at 2 Hours Post-dose
Description: Absence or presence of phonophobia was recorded by the participants on a paper diary. Absence is defined as no phonophobia at 2 hours post-dose.
Time Frame: 2 hours post-dose
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg ODT | Placebo
Number analyzed (Participants) | 92 | 96
Participants | 72 | 55

6. Secondary Outcome: Number of Participants With Absence of Nausea at 2 Hours Post-dose
Description: Absence or presence of nausea was recorded by the participants on a paper diary. Absence is defined as no nausea at 2 hours post-dose.
Time Frame: 2 hours post-dose
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg ODT | Placebo
Number analyzed (Participants) | 92 | 96
Participants | 82 | 73

7. Secondary Outcome: Number of Participants With Absence of Functional Disability at 2 Hours Post-Dose
Description: Level of functional disability was assessed on a paper diary by the participants.
  Level of functional disability was rated as: normal, mildly impaired, severely impaired or unable to do activities, requires bed rest. Absence of functional disability defined as a rating of normal at 2 hours post-dose.
Time Frame: 2 hours post-dose
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Rizatriptan 10 mg ODT | Placebo
Number analyzed (Participants) | 92 | 96
Participants | 66 | 42

ADVERSE EVENTS:
Arm/Group | Rizatriptan 10 mg ODT | Placebo
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/96
Other Adverse Events (participants affected / at risk) | 6/92 | 3/96
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rizatriptan 10 mg ODT (N=92) | Placebo (N=96)
Hyperchlorhydria (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Feeling cold (General disorders) | 0 | 1
Feeling jittery (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
In the Adverse Events section, all non-serious adverse experiences reported are post-treatment, up to the time of taking rescue medication or 14 days post-dose, whichever comes first.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.